CLINICAL TRIAL: NCT06314581
Title: Effect of a Multifaceted Educational Intervention on the Implementation of Evidence-based Practices for Benign Paroxysmal Positional Vertigo in an Emergency Department
Acronym: BPPV-Teaching
Status: Active, not recruiting | Type: Observational
Sponsor: Fondation Hôpital Saint-Joseph (Other)
Responsible Party: Sponsor
Other Study IDs: 673_BPPV-Teaching
Record Dates: First submitted 2024-03-11; First posted 2024-03-18 (Actual); Last update posted 2024-05-30 (Actual); Status verified 2024-05

CONDITIONS: Benign Paroxysmal Positional Vertigo
MeSH Terms: conditions — Benign Paroxysmal Positional Vertigo

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- BPPV

SUMMARY:
Acute vertigo accounts for around 4% of emergency room visits. Triggered episodic vestibular syndrome is the most commonly encountered symptomatic context. BPPV (Benign Paroxysmal Positional Vertigo) is the main cause, representing 40-50% of the vertigo cases assessed in emergency departments. It results from the migration of calcium carbonate particles (otoliths), from the sticky membrane of the utricle and saccule of the inner ear, to one of the 3 semicircular canals (SCC), posterior, horizontal or lateral, and anterior. It occurs idiopathically with head movement, through degeneration, or following head trauma. The otolith impulse causes the endolymph to move, temporarily and aberrantly displacing the cup of the affected canal, resulting in the transmission of erroneous information to the vestibular nuclei. This leads to the sudden onset of vertigo and eye deviation, resulting in transient nystagmus. The location of the displaced otoliths determines the variant of BPPV: BPPV of the posterior semicircular canal is the most common (around 65% of BPPVs), followed by BPPV of the horizontal canal, while BPPV of the anterior canal is rare, as it resolves spontaneously and rapidly. Although a benign condition, BPPV leads 9 times out of 10 to a medical consultation, interruption of daily activities, or sick leave. Untreated, it will usually recur, and can impact on patients' quality of life.

DETAILED DESCRIPTION:
Recommendations for the appropriate management of vertigo in emergency departments published in 2023 reaffirmed that the management of BPPV is based solely on the clinic. There is no imaging test that can confirm the presence of otoliths migrating to a semicircular canal during head movement. BPPV should be suspected in the presence of an episodic vestibular syndrome triggered by head movements, and more broadly, in the presence of brief vertigo without a clear cause and without spontaneous or lateral facing nystagmus. The diagnosis of posterior BPPV is made when vertigo is accompanied by transient vertical torsional nystagmus on the Dix-Hallpike test. In some cases of BPPV, the Dix-Hallpike test produces vertigo, but not transient nystagmus. This phenomenon is known as "subjective BPPV", and may affect up to a quarter of patients suspected of having BPPV. It can be explained by a low otolith load in the affected canal, by spontaneous healing by otolith egress from the canal , but also by poor technique on the part of the clinician (slow maneuver or faulty final position). In patients with a typically positive Dix-Hallpike result or subjective BPPV, 1st-line treatment is based on a canalith repositioning maneuver. The modified Epley maneuver is the recommended one, and its efficacy is supported by numerous meta-analyses. It is significantly associated with complete resolution of symptoms after 7 days. Horizontal BPPV should be suspected by the presence of transient horizontal nystagmus in the Dix-Hallpike test. The Supine Head Roll test then confirms the diagnosis, with the appearance of vertigo and transient horizontal geo- or ageo-tropic nystagmus. The preferred treatment maneuver is Lempert's "Barbecue" maneuver. This management strategy can be summarized in a decision tree. As posterior BPPV is the most common, the appropriate use of the Dix-Hallpike and Epley maneuvers has a positive effect on a large majority of BPPV patients in emergency departments In terms of clinical decision rules, the management of vertigo has been mentioned as the 1st priority of emergency physicians . However, numerous studies have highlighted the fact that their clinical approach is often inappropriate and leads to underdiagnosis of BPPV. Under-diagnosis is generally due to failure to verify the existence of spontaneous nystagmus, under-use of the Dix-Hallpike test, or its misuse. While BPPV is a common and easily treatable condition, its diagnosis and treatment are largely delayed by a lack of theoretical knowledge and clinical skills among physicians.

Understanding the orientation of the vestibular apparatus and how it is stimulated is difficult learning. Traditional lecture-based learning appears to have little gain in terms of skill acquisition. This approach is tedious and offers little opportunity to acquire clinical skills. Theoretical resources do exist; in particular, the BPPV Viewer software, which offers 3D modeling of the vestibular apparatus, and the demonstration videos by Prof. Peter Johns available on Youtube® could provide a fairly clear theoretical basis. Proposing new teaching methods could be one way of solving the problem of sub-optimal management of BPPV and the resulting under-diagnosis. Two original teaching methods have been published, one using demonstrations involving students to teach vestibular physiology, the other based on Gagne's 9 event. The retention and transfer of knowledge to the bedside needs to be investigated.

ELIGIBILITY:
Inclusion Criteria:

* age >18
* A triggered episodic vestibular syndrome defined by vertigo that may be associated with nausea or vomiting, brief (< 1 minute) and transient, triggered by changes in head or body position;
* Or brief episodes of vertigo with no obvious cause and no spontaneous nystagmus.
* French speaking

Exclusion Criteria:

* Existence of one or more BPPV diagnostic non-compliance criteria i.e. impaired alertness (Glasgow Coma Score <15), nystagmus present in spontaneous or lateral gaze (without or with Frenzel glasses), headache or neck pain, hypoacusis concomitant with vertigo, any central neurological sign, otalgia, tinnitus, alcohol intoxication;
* Existence of one or more contraindications to performing the Dix-Hallpike test, i.e. vertebro-basilar insufficiency, recent fracture or dislocation of a cervical vertebra, cervical arthritis, recent cervical surgery, history of sino-carotid syncope;
* Patient under court protection;
* Patient under guardianship or curatorship;
* Patient deprived of liberty;
* Patients who object to the use of their data.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient older than 18 , visiting the emergency room for vertigo
Sampling Method: Non-Probability Sample
Enrollment: 382 (Actual)
Dates: Start 2023-05-01 (Actual); Primary Completion 2024-05-01 (Actual); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
accurate BPPV diagnostics | one year
  Percentage of appropriate BPPV diagnoses, i.e., positive diagnostic tests obtained with eligible patients, before and after the educational intervention.
  Positive diagnostic tests for BPPV are defined as follows:
  * A Dix-Hallpike test producing triggered and transient, vertical and torsional nystagmus or isolated transient and paroxysmal vertigo (subjective BPPV) on the affected side for the appropriate diagnosis of posterior BPPV,
  * A Supine Head Roll test producing a triggered and transient horizontal, geotropic or agiotropic nystagmus observed on both sides, but more intense on the healthy side, for the appropriate diagnosis of horizontal BPPV.

SECONDARY OUTCOMES:
therapeutic maneuvers performed | 1 year
  Percentage of therapeutic maneuvers performed (Epley and Barbecue, respectively) by trained clinicians on patients with a positive diagnostic test for BPPV, before and after the educational intervention.
Satisfaction of clinicians who received the educational interventio | one year
  Satisfaction of clinicians who received the educational intervention at the end of their clinical management, assessed on a 5-point Likert scale.

CONTACTS AND LOCATIONS:
Locations (1):
- Groupe Hospitalier Paris Saint-Joseph, Paris, France